CLINICAL TRIAL: NCT04621006
Title: The Contact Activation System and Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: UMC Utrecht (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Morten Lee Halling, Principal Investigator, Esbjerg Hospital - University Hospital of Southern Denmark
Other Study IDs: CAS UC
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis
Keywords: Misfolded protein; Coagulation Factor XII; Kallikrein; High Molecular Weight Kininogen; The contact activation system; Endoplasmatic reticulum stress; Misfolded alpha-1-antitrypsin; Inflammatory bowel disease; Inflammation
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma (EDTA and citrate) stored at -70 degrees celcius. Fecal extract stored at -70 degrees celcius. Colonic tissue snap frozen with liquid nitrogen and stored at -70 degrees celcius.
  Colonic tissue fixated in formalin and embeded in parafin within 72h.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UC group: Patients with active ulcerative colitis
  Interventions: Diagnostic Test: Continuously assessment of disease activity

INTERVENTIONS:
Diagnostic Test: Continuously assessment of disease activity — Continuous measures of disease activity and activity in the contact activation system.

SUMMARY:
The study aims to describe alterations in the contact activation system during active and inactive ulcerative colitis.

Contact activation system measures are compared in a cross sectional (healthy controls vs. active disease) and longitudinal (active diasese vs. inactive disease) fashion.

DETAILED DESCRIPTION:
We include and follow up on 102 adults with active ulcerative colitis. Visits are week 0 (inclusion), 6, 12 and 26 (end of study). We obtain plasma and fecal samples at each visit. Whereas we obtain colonic tissue samples only at inclusion and end of study.

Registered data are:

* Demographics realate to UC and general wellbeing.
* Clinical parametres used for UC evaluation are PRO2, SCCAI, CRP, fecal calprotectin, Mayo endoscopic subscore and Nancy index.
* The contact activation system is characterised by FXII, prekallikrein, kallikrein generation, HK, cHK (specific to plasma kallikrein), cHK (specific to tissue kallikrein), C1 inhibitor and Kallistatin.
* Polymerized alpha-1-antitrypsin is characterised by the degree of polymerization and the capacity to activate the contact activation system.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill diagnostic criteria of ulcerative colitis
* SCCAI score ≥ 5
* Mayo Endoscopic Subscore ≥ 1
* Age ≥ 18 years
* Most understand written and oral information in Danish
* Informed consent must be given

Exclusion Criteria:

* Pregnancy
* Infection at inclusion
* Any existing disease at inclusion:

  * liver disease or defect in CAS
  * inflammatory rheumatologic or dermatologic disease
  * cardiovascular or renal disease
  * immunodeficiency or hematologic diseases
  * malignancies
* Medication with

  * Systemic corticosteroids at inclusion
  * ACE-inhibitor
  * Acetylsalicylic acid/NSAID
  * Warfarin, Phenprocoumon, NOAC and heparins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled from the Department of Medical Gastroenterology at the Hospital of Southwest Jutland, Region of Southern Denmark, Denmark
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical disease activity. | End of study (August 28th, 2024)
  PRO2 score, 0-6 points. A score of one or more defines active disease.
Endoscopic disease activity. | End of study (August 28th, 2024)
  Mayo endoscopic score, 0-3 points. A score of one or more defines active disease.
Kallikrein generation | End of study (August 28th, 2024)
  The assay reflects the downstream activation of the contact activation system which allows us to determine the amount of kallikrein generated in each sample.
Polymerised alpha-1-antitrypsin in participants | End of study (August 28th, 2024)
  A Western blot verifies the present of polymerised alpha-1-antitrypsin.
Polymerised alpha-1-antitrypsin as an activator of the contact activation system | End of study (August 28th, 2024)
  We add polymerised alpha-1-antitrypsin to our kallikrein generation. If kallikrein is generated the polymers activated the system.
Localisation of contact activation system components in tissue samples | End of study (August 28th, 2024)
  Immunhistochemical methods locate FXII, PK, cHK (specific to plasma kallikrein and tissue kallikrein), C1 Inhibitor, and Kallistatin in biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Morten L Halling, M.D., Principal Investigator — Department of Medical Gastroenterology, University Hospital of Southern Denmark - Esbjerg
Locations (1):
- Department of Medical Gastroenterology, University Hospital of Southern Denmark, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No